CLINICAL TRIAL: NCT01949038
Title: Comparison Between Sublingual and Oral Alprazolam as Conscious Sedation for Upper Gastrointestinal Endoscopy
Brief Title: Alprazolam as Conscious Sedation for Upper Gastrointestinal Endoscopy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Gholamrezaei, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 391009
Record Dates: First submitted 2013-09-17; First posted 2013-09-24 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Diagnostic Esophagogastroduodenoscopy
Keywords: Pain; Discomfort; Anxiety; Satisfaction; Compliance
MeSH Terms: conditions — Pain; Anxiety Disorders; Personal Satisfaction; Patient Compliance | interventions — Alprazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oral placebo (Placebo Comparator): Patients receive one oral dose of placebo least 30 minutes before the procedure.
  Interventions: Drug: Oral placebo
- Sublingual placebo (Placebo Comparator): Patients receive one oral dose of placebo at least 30 minutes before the procedure.
  Interventions: Drug: Sublingual placebo
- Sublingual alprazolam (Active Comparator): Patients receive one oral dose of alprazolam 0.5 mg at least 30 minutes before the procedure.
  Interventions: Drug: Sublingual alprazolam
- Oral alprazolam (Active Comparator): Patients receive one oral dose of alprazolam 0.5 mg at least 30 minutes before the procedure.
  Interventions: Drug: Oral alprazolam

INTERVENTIONS:
Drug: Oral alprazolam
  Arms: Oral alprazolam
Drug: Sublingual alprazolam
  Arms: Sublingual alprazolam
Drug: Oral placebo
  Arms: Oral placebo
Drug: Sublingual placebo
  Arms: Sublingual placebo

SUMMARY:
Diagnostic esophagogastroduodenoscopy is an uncomfortable and stressful procedure for most of the patients. Various methods are available for sedation during this procedure. Because of some side effects related to intravenous administration of sedatives, oral administration of these drugs is under attention. Alprazolam is a benzodiazepine which is used mainly in treatment of anxiety. Hence, we determine the efficacy of oral and sublingual alprazolam as for sedation during this procedure. We hypothesize that sublingual alprazolam is more effective than that oral form and both forms more effective than placebo in reducing anxiety and pain/discomfort related to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Referring for upper GI endoscopy
* Age 18 to 65 years
* First experience of upper GI endoscopy
* Class I or II of American Anesthesiology Association
* Willingness to participate

Exclusion Criteria:

* Severe psychiatric, neurological, cardio-vascular, or renal disorders
* History of allergy or intolerance to benzodiazepines or lidocaine
* History of upper GI surgery
* Pregnancy or lactation
* GI anomalia during endoscopy
* Need for therapeutic procedures during endoscopy
* Active bleeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Procedure related pain/discomfort | Within the first one hour after the procedure
  Procedure related pain/discomfort is assessed by patients on a 11-point numeric rating scales after the procedure.

SECONDARY OUTCOMES:
Pre-procedure anxiety | Before and 30 minutes after medication
  Procedure related anxiety is assessed by patients on a 11-point numeric rating scales before and 30 minutes after the medication.
Patients' satisfaction | Within the first one hour after the procedure
  Procedure related patients' satisfaction is assessed by patients on a 11-point numeric rating scales after the procedure.
Compliance | Within the first one hour after the procedure
  Compliance is assessed by patients from no compliance (0) to excellent compliance (4) after the procedure.
Duration of the procedure | Within the first one hour after the procedure
  Duration of the procedure is recorded.
Side effects | Within the first one hour after the procedure
  Any side effects attributed to alprazolam is assessed Within the first one hour after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Shavakhi, M.D., Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Private Outpatient Clinic of Gastroenterology, Isfahan, Isfahan, Iran

REFERENCES:
- [Background] Hedenbro JL, Ekelund M, Aberg T, Lindblom A. Oral sedation for diagnostic upper endoscopy. Endoscopy. 1991 Jan;23(1):8-10. doi: 10.1055/s-2007-1010598. PMID 2009843
- [Derived] Shavakhi A, Soleiman S, Gholamrezaei A, Khodadoostan M, Shavakhi S, Tahery A, Minakari M. Premedication with sublingual or oral alprazolam in adults undergoing diagnostic upper gastrointestinal endoscopy. Endoscopy. 2014 Aug;46(8):633-9. doi: 10.1055/s-0034-1377305. Epub 2014 Jun 30. PMID 24977401